CLINICAL TRIAL: NCT03100279
Title: Psychotherapy Process and Outcomes in Cognitive-Behavioral Treatment for Anxious and Depressed Youth
Brief Title: Process and Outcomes in CBT for Anxious and Depressed Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers University (Other)
Responsible Party: Principal Investigator, Brian Chu, Associate Professor, Rutgers University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-504Rc11
Record Dates: First submitted 2017-03-14; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Anxiety Disorders; Depression
Keywords: cognitive behavioral therapy; treatment mediators; trajectories of change
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: This study will employ a quasi-experimental open-trial design that includes a comprehensive diagnostic assessments at pre- and post-treatment (diagnostic interview, symptom and functioning measures, and prospective mediators) and continuous assessment throughout an active treatment phase. Anxiety/depression symptoms will be assessed each session and prospective mediators (cognitive, behavioral, and affective variables) will be assessed every four sessions. A two-week baseline period will separate the initial intake from the first treatment session. The traditional ABAB experimental single-case design will not be used because it is not appropriate in clinical situations where the removal of treatment intervention could be harmful to clinical patients (Kazdin, 1992). Each youth who meets inclusion criteria will complete a two-week baseline phase that includes three assessments (intake, phone follow-up, and first session).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT for Anxiety or Depression (Experimental): If a youth meets criteria for a primary diagnosis of clinical or subclinical depressive disorder she or he will be assigned to Primary and Secondary Control Enhancement Therapy (PASCET; Weisz et al., 1987). If a youth meets criteria for a primary diagnosis for a clinical or subclinical anxiety disorder, she or he will be assigned to the Coping Cat (Kendall, 2000). Both CBT treatments include a therapist manual and companion workbooks for the youth. CBT teaches coping skills that help anxious and depressed youth challenge anxious and depressive thinking. It also helps the child habituate to negative physiological feelings and learn skills to cope with emotional distress.
  Interventions: Behavioral: Coping Cat/CAT Project; Behavioral: Primary and Secondary Coping Enhancement Therapy

INTERVENTIONS:
Behavioral: Coping Cat/CAT Project — The "Coping Cat" program, developed by Kendall and colleagues (Kendall, 1994; Kendall, 2000; Kendall, Kane, Howard, & Siqueland, 1989; Kendall, Flannery-Schroeder et al., 1997), involves (1) teaching children to identify their own anxious feelings and physiological signs of anxiety, (2) teaching children to identify their own anxiety-provoking cognitions, (3) developing a plan to guide coping - a plan that involves changing the child's thoughts (into positive self-talk) and actions (into self-initiated exposures), and (4) self-evaluation and self-reward. The therapist uses modeling (e.g., revealing therapist's own anxiety and sharing successful coping experiences), in vivo exposure tasks, role-playing (e.g., to prepare for exposure tasks), relaxation training, and contingent reinforcement (e.g., for trying and for succeeding at exposure tasks), in developing these four themes.
Behavioral: Primary and Secondary Coping Enhancement Therapy — PASCET is a brief (11-15 sessions) CBT program for depressed youths typically aged 8-15. Sessions and practice assignments are built on findings concerning cognitive and behavioral features of youth depression (e.g., Lewinsohn et al., 1990; Stark et al., 1987), and on the two-process model of perceived control and coping (Rothbaum, Weisz, & Snyder, 1982; Weisz et al., 1984a,b). In this model, primary control involves efforts to cope by making objective conditions (e.g., one's activities, one's peer status) conform to one's wishes. In contrast, secondary control involves coping by adjusting oneself (e.g., one's expectations, interpretations) to fit objective conditions, so as to influence their subjective impact without altering the actual conditions. The goal is for youngsters to build their skills in primary and secondary control coping, and apply those skills to events and conditions that can trigger depression. Therapists are guided by a Therapist's Manual and use a youth workbook.

SUMMARY:
The current study will evaluate the predictors, mediators, outcomes, and critical therapy processes associated with manual-based psychological therapies for 400 youth (ages 7-16 years) with anxiety and/or depression seeking services within a semi-natural clinic setting. Essentially, this study seeks to determine "what works" about psychological therapy for youth.

DETAILED DESCRIPTION:
The current study will evaluate the efficacy of manual-based psychological therapies administered with youth with anxiety and mood problems. It will also assess the role of several mediators (e.g., coping skills, negative self-statements, parenting practices) hypothesized to maintain youth anxiety and depression. Youth (ages 7 - 16) diagnosed with a principal Anxiety or Depressive Disorder will be recruited to receive Cognitive-Behavioral Therapy (CBT). Anxiety (e.g., Generalized Anxiety Disorder, Separation Anxiety Disorder, Social Phobia) and depressive disorders (e.g., Major Depression Disorder, Dysthymia Disorder) are among the most common emotional disorder affecting America's youth, with 12-20% of youth meeting criteria for an anxiety disorder and 2-5% meeting criteria for depression at any one point in time. Both forms of disorders are associated with significant distress and functional impairment in school, peer, and family domains. Left untreated, early affliction with these disorders leaves individuals at risk for adult anxiety disorders, chronic depression, substance abuse, and long-term functional impairment. Identifying efficacious treatments and their most effective, "active ingredients" is a top health research priority. In addition, knowledge about how our psychotherapies work lags behind research documenting simple treatment effects. Knowing the therapy techniques that have the best outcomes as well as knowing how those interventions produce gains will provide valuable information for improving our already effective therapies.

Two manual-based psychological treatments that have received empirical support in clinical trial outcome studies are cognitive-behavioral treatment for anxious children (Kendall's Coping Cat) and cognitive-behavioral treatment for depressed children (Weisz's PASCET). Both treatments (a) use a manual and (b) have been supported in clinical trial outcome studies where youth receiving the manualized treatment interventions improve more than the control groups. The Kendall treatment program has produced some of the strongest treatment effects yet seen in the empirical literature for children and adolescents.

Despite our increasing knowledge of treatments that work, there has been insufficient analysis of psychological mediators in youth psychotherapy. Research on psychological mediators, or "mechanisms of action," provide information about how psychotherapy works. Randomized clinical trials document that CBT produces clinical outcomes, such as decreased symptoms and impairment following treatment. Fewer studies have assessed the degree to which coping skills, emotion management, or cognitive restructuring mediate these clinical gains. This type of mediator analysis is essential to test the theory underlying our treatments and helps inform our models of pathology. For example, if increased primary (active) coping skills precede a reduction in depressive symptoms, we might infer that poor coping skills are a maintaining factor of depression and that successful therapy works by increasing a youth's use of such skills.

In the current study, we will invite youth to participate in a CBT intervention with demonstrated efficacy and will conduct a thorough assessment of potential therapy process and mediator variables that impact treatment outcomes. Both primary (active problem solving) and secondary (attempts to adjust to situations that can not be changed) coping skills have been linked to a number of psychological distress states in youth and may have specific links to maintaining depression in youth. In anxious youth, the ratio of negative to positive self-talk has been shown to mediate gains in CBT. The role of parenting practices has also been highlighted as an important maintaining factor in anxiety (e.g., modeled anxious behavior, parent intrusiveness). Self-efficacy, a cognitive appraisal of one's ability to manage challenges, has also been related to distress in youth. Affective components, such as positive affect, negative affect, and physiological hyperarousal have received increased attention because of they reflect basic emotional processes that underlie and distinguish anxiety and depressive disorders. Finally, less research has identified cognitive functioning related to anxiety and depression, but experts encourage the assessment of multidimensional cognitive factors in the expression of psychological distress to enhance our ability to factor in normative developmental processes. Given this, the current study will assess youth primary and secondary coping skills, youth automatic thoughts and self-statements, parenting practices, affective processes and cognitive functioning as treatment outcomes and potential mediators of symptom change in CBT.

There have also only been minimal attempts to explore the therapist and client factors that impact within-session therapy processes that could improve the delivery of our empirically-supported treatments. Process factors like client engagement and therapeutic alliance may deserve particular attention in youth-based therapies because youth rarely refer themselves for treatment, often do not recognize or acknowledge the existence of problems, and frequently are at odds with their parents about the goals of therapy. Recent empirical data suggests that youth demonstrating greater engagement or stronger therapeutic alliance may experience better treatment outcomes. Therapist responsiveness to child needs and flexibility in implementing manual-based therapies might also have significant, if indirect, effects on successful treatment. A greater understanding of therapist, child, and interpersonal factors that improve the delivery of therapy could lead to concrete recommendations in training novice clinicians or in developing improved versions of current therapy manuals.

Because treatment will occur within a semi-natural clinic setting, a multiple baseline, single-case design will be used. Employing a single-case design in this context will permit continuous assessment throughout baseline and treatment phases. This design will provide data for the course and sequence of symptom and mediator change. We will also be able to document the sequence of symptom change as it relates to the introduction of specific treatment interventions. The combined information can provide valuable information for how these treatments work and which interventions produce what specific client change.

II. SPECIFIC AIMS

The current study will attempt to address the following aims:

Aim 1. Determine whether CBT for anxiety and depression are effective in a natural clinic setting where cases exhibit greater range of symptom severity, multiple clinical problems, and greater socioeconomic and cultural diversity. Effectiveness will be assessed in diagnostic, symptom, and adaptive functioning domains, including executive cognitive functioning.

Aim 2. Determine if youth coping skills, behavioral activation, automatic thoughts, affective process, self-efficacy or parenting practices mediate the relationship between CBT interventions and clinical outcomes.

Aim 3. Determine if youth or therapist within-session processes (e.g., child involvement, therapeutic alliance, therapist adherence to treatment protocol) moderates treatment success.

Aim 4. Determine the pattern of symptom change associated with CBT for youth (e.g., gradual symptom decline, presence of sudden gains).

Aim 5. Note patterns of additional youth mental health services and auxiliary services that families seek beyond treatment received at the Youth Anxiety and Depression Clinic.

ELIGIBILITY:
Inclusion Criteria:

We expect 200 youth (ages 7-16 years) with a primary anxiety disorder and 200 youth (ages 7 - 16 years) with a primary depressive disorder to serve as participants. To participate, a youth must meet criteria for a primary DSM-IV-TR (American Psychiatric Association, 2000) diagnosis of Generalized Anxiety Disorder, Separation Anxiety Disorder, Social Phobia, Specific Phobia, Panic Disorder with or without a history of Agoraphobia, Major Depression Disorder, Minor Depression, or Dysthymia. Diagnosis will be based on both youth and parent report during an Independent Evaluator (IE) semi-structured interview. Youth may also participate with a subclinical diagnosis for any of these disorders if: (a) the youth demonstrates sufficient symptoms but does not yet reach clinical levels of impairment OR (b) the youth demonstrates only several symptoms related to the above disorders but demonstrates clinical impairment, AND (c) the consenting parent agrees that anxiety or mood problems would be appropriate as a clinical focus for treatment. Allowing youth with subclinical diagnoses will allow the study to investigate the effectiveness of the therapies across a range of clinical severity. This design models usual community care where a larger range of severity is witnessed and many youth may not meet all criteria for formal diagnosis. After receiving an initial diagnostic assessment, the parent must consent and the youth must assent to continued participation in the study and must be willing to receive psychological therapy at the Youth Anxiety and Depression Clinic (YAD-C), a specialty program within the outpatient clinic of the Rutgers University Graduate School of Applied and Professional Psychology (GSAPP).

Exclusion Criteria:

Youth who have a primary diagnosis of a DSM-IV disorder other than anxiety or depression (e.g., anorexia nervosa, Postraumatic Stress Disorder, Attention Deficit-Hyperactivity Disorder), or who have received any diagnosis of mental retardation, a pervasive developmental disorder, schizophrenia, or bipolar disorder will be excluded. Youth who demonstrate suicidal ideation or intent (by child or parent report) severe enough to require current hospitalization, or youth who have attempted suicide in the past 3 months, will also be excluded. These clinical problems require specialized treatment that YAD-C is not prepared to offer.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2005-07-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Global Impression - Severity (CGI-S) Scale: interviewer | Change from pre-treatment to post-treatment (an average of 16 weeks)
  The CGI-S score provides a global rating of baseline severity ranging from 1 (not at all ill) to 7 (extremely ill). The IE will provide a baseline CGI ratings for each patient at pretreatment and posttreatment.

SECONDARY OUTCOMES:
Change in Anxiety Disorders Interview Schedule (ADIS-IV) - Principal Diagnosis | Change from pre-treatment to post-treatment (an average of 16 weeks)
  The ADIS-C/P (Silverman & Albano, 1996) is a semi-structured interview consisting of independent but comparable parent and child interviews that have good interviewer reliability (e.g., k= .98, parent interview; k=.93, child interview; Silverman & Nelles, 1988), retest reliability (i.e., r=.76, parent interview; Silverman & Eisen, 1992), and sensitivity to treatment effects (e.g., Albano, Know, & Barlow, 1995; Kendall et al., 1997). The parent and child interviews are conducted individually allowing the diagnostician to derive parent-reported, child-reported, and composite (parent and child) diagnoses. Diagnosticians will be trained to reliability by shadowing trained interviewers, being shadowed by a trained interviewer, and by coding videotaped interviews and matching gold-standard ratings of diagnoses.
Change in Children's Depression Rating Scale-Revised (CDRS-R): Total depression score | Change from pre-treatment to post-treatment (an average of 16 weeks)
  Clinicians rate 17 symptom areas covering academic, social, health and cognitive functioning. Administered alone, the CDRS-R takes 15-20 minutes to complete. Administered with the ADIS-IV, it requires an additional 5 minutes with the parent or child because many questions overlap. The majority of ratings also get completed by the Interviewer after the ADIS is completed (not directly with parent or child).
Change in Strengths and Difficulties Questionnaire total impairment - parent report | Change from pre-treatment to post-treatment (an average of 16 weeks)
  a brief 25-item behavioral screening questionnaire assessing 5 domains (emotional symptoms, conduct problems, hyperactivity/inattention, peer relationships problems, and prosocial behaviors). Parents and youth will rate this at pre- and posttreatment.
Change in Strengths and Difficulties Questionnaire total impairment - child report | Change from pre-treatment to post-treatment (an average of 16 weeks)
  a brief 25-item behavioral screening questionnaire assessing 5 domains (emotional symptoms, conduct problems, hyperactivity/inattention, peer relationships problems, and prosocial behaviors). Parents and youth will rate this at pre- and posttreatment.
Change in State-Trait Anxiety Inventory for Children (STAIC) - Trait Scale: parent | Trajectory of change across weekly sessions (weeks 1 through completion; on average 16 weeks)
  The STAIC-Trait scale (Speilberger et al., 1973) is a 20-item scale that assesses global anxiety that remains consistent across situations (trait anxiety). Only youth will complete this measure. Normative and reliability data are available (Spielberger et al., 1973). Factor-analytic studies support the state-trait distinction (Finch, Kendall, & Montgomery, 1974).
Change in State-Trait Anxiety Inventory for Children (STAIC) - Trait Scale: child | Trajectory of change across weekly sessions (weeks 1 through completion; on average 16 weeks)
  The STAIC-Trait scale (Speilberger et al., 1973) is a 20-item scale that assesses global anxiety that remains consistent across situations (trait anxiety). Only youth will complete this measure. Normative and reliability data are available (Spielberger et al., 1973). Factor-analytic studies support the state-trait distinction (Finch, Kendall, & Montgomery, 1974).
Change in Revised Children's Anxiety and Depression Scale (RCADS) - Parent | Change from pre-treatment to post-treatment (an average of 16 weeks)
  RCADS-C/P (Chorpita, Yim, Moffitt, Umemoto,& Francis, 2000) is a 47-item scale whose items correspond closely to DSM-IV anxiety and major depressive disorders. Parallel parent and child versions will be used. Factor analysis has yielded subscales associated with the diagnoses of interest (e.g., Separation Anxiety Disorder, Social Phobia, Generalized Anxiety Disorder, Major Depressive Disorder). The subscales demonstrated good factorial validity, internal consistency, one-week test-retest reliability, and good convergent and discriminant validity (Chorpita et al., 2000). It has also demonstrated reasonable convergent validity with other leading anxiety and depression measures (e.g., Revised Children's Manifest Anxiety Scale, Children's Depression Inventory; Chorpita et al., 2000). The RCADS-Parent Form (RCADS-P) is a 47-item parent-report version of the youth RCADS.
Change in Revised Children's Anxiety and Depression Scale (RCADS) - depression subscale | Trajectory of change across weekly sessions (weeks 1 through completion; on average 16 weeks)
  The depression subscale is the 10-items from the long form that assesses depression symptoms.
Change in Multidimensional Anxiety Scale for Children - Child | Change from pre-treatment to post-treatment (an average of 16 weeks)
  Multidimensional Anxiety Scale for Children - Child and Parent Forms (March, 1997). The MASC includes both a long form (39-items) and a short form (10-items; MASC-10) designed for repeated assessments. Parallel parent and child versions will be used. The long form consists of 39 items, rated on a "0" (Never True) to "3" (Often True about me) scale, distributed across four broad scales (Physical Symptoms, Harm Avoidance, Social Anxiety, Separation/Panic) that also has six subscales. The MASC has been normed on large samples and is one of the most widely used anxiety symptom measures. The 10-item short form (MASC-10) can be administered rapidly (1 min) for repeated testing.
Change in Multidimensional Anxiety Scale for Children - Parent | Change from pre-treatment to post-treatment (an average of 16 weeks)
  Multidimensional Anxiety Scale for Children - Child and Parent Forms (March, 1997). The MASC includes both a long form (39-items) and a short form (10-items; MASC-10) designed for repeated assessments. Parallel parent and child versions will be used. The long form consists of 39 items, rated on a "0" (Never True) to "3" (Often True about me) scale, distributed across four broad scales (Physical Symptoms, Harm Avoidance, Social Anxiety, Separation/Panic) that also has six subscales. The MASC has been normed on large samples and is one of the most widely used anxiety symptom measures. The 10-item short form (MASC-10) can be administered rapidly (1 min) for repeated testing.
Change in Multidimensional Anxiety Scale for Children - Brief form | Trajectory of change across weekly sessions (weeks 1 through completion; on average 16 weeks)
  This is the 10-item brief form of the MASC.
Change in Center for Epidemiologic Studies-Depression Scale (CES-D) - Child | Change from pre-treatment to post-treatment (an average of 16 weeks)
  The CES-D (parent and child forms) includes 20 items designed to assess depressed mood, feelings of worthlessness/guilt, sense of helplessness/hopelessness, psychomotor retardation, loss of appetite, and sleep disturbance. Parallel parent and child versions will be used. Using a four-point scale, respondents indicate the frequency with which symptoms have been experienced during the past week. Response categories include 0 = rarely (less than 1 day); 1 = little (1-2 days); 2 = moderately (3 to 4 days); or 3 = most of the time (5-7 days). Four items are reverse-scored, and a composite is calculated by summing item responses (range 0-60). CES-D was developed with adults but has been applied without adaptation to young adolescents. A cutoff point of 16 and above for screening adolescents for current major depressive disorder or dysthymia is considered optimal.
Change in Center for Epidemiologic Studies-Depression Scale (CES-D) - Parent | Change from pre-treatment to post-treatment (an average of 16 weeks)
  The CES-D (parent and child forms) includes 20 items designed to assess depressed mood, feelings of worthlessness/guilt, sense of helplessness/hopelessness, psychomotor retardation, loss of appetite, and sleep disturbance. Parallel parent and child versions will be used. Using a four-point scale, respondents indicate the frequency with which symptoms have been experienced during the past week. Response categories include 0 = rarely (less than 1 day); 1 = little (1-2 days); 2 = moderately (3 to 4 days); or 3 = most of the time (5-7 days). Four items are reverse-scored, and a composite is calculated by summing item responses (range 0-60). CES-D was developed with adults but has been applied without adaptation to young adolescents. A cutoff point of 16 and above for screening adolescents for current major depressive disorder or dysthymia is considered optimal.
Change in Adolescent Alcohol and Drug Involvement Scale (AADIS): incidents of substance abuse | Change from pre-treatment to post-treatment (an average of 16 weeks)
  For youth 13 years and older, diagnosticians will complete the Adolescent Alcohol and Drug Involvement Scale (AADIS) to screen for alcohol and substance use. All teens will be asked if they have ever used tobacco, alcohol, or marijuana and then interviewers will give a general prompt for other substance use. If the teen endorses use of other elicit or controlled substances, frequency ratings will be obtained. If the teen endorses any substance use, the interviewer will administer an additional 14 items assessing the context, function, and history of drug and alcohol use. The AADIS has been tested to be reliable and appropriate for adolescent respondents (Winters, 2003).
Change in Olweus Bully/Victim Questionnaire - Parent and Child report (OBVQ-P/C): frequency of victimization events | Change from pre-treatment to post-treatment (an average of 16 weeks)
  The OBVQ (Solberg & Olweus, 2003), designed for grades 3-10, is used to assess experiences with being bullied and bullying others. The OBVQ will be administered as an interview, individually with the child and parent/s, following the other clinician-administered measures (ADIS, AADIS, SACA). A shortened and revised version of the original OBVQ (28 items) will be used that includes global assessment of being bullied and bullying others, as well as specific items that assess nine different forms of bullying including hitting and kicking, spreading false rumors, ignoring peers, and bullying of a sexual or racial nature. The OBVQ demonstrated adequate internal consistency (alpha > .80), and construct and criterion-related validity have been reported (Solberg & Olweus, 2003).
Change in Multidimensional Bullying Impact Scale (MBIS) - total impairment score | Change from pre-treatment to post-treatment (an average of 16 weeks)
  The MBIS is a recently developed measure (Chu, B. C., Hoffman, L., Johns, A., Reyes-Portillo, J., & Hansford, A, 2014) that assesses socio-emotional impairment related to bullying in school-aged youth. The BIS is a 44-item measure, rated 0 (not at all) to 3 (most of the time; total range: 0 - 60). Initial piloting demonstrated that BIS total scores correlated with bullying experiences and anxiety and depressive symptoms (Chu et al., 2014). Items begin with the clause, "When I have been bullied, I..." and assess the frequency that victimization negatively impacts family relations, peer relations, academic performance and attendance, and extracurricular participation.
Change in Child Behavior Checklist (CBCL) - total internalizing score | Change from pre-treatment to post-treatment (an average of 16 weeks)
  The CBCL (Achenbach, 2001) is a 118-item parent-report scale assessing behavioral problems and social competencies. Only parents will complete this measure. Items are rated from not true (0) to very true or often true (2). The CBCL has broadband internalizing and externalizing factors and eight specific scales (e;g., anxiety-depression). Normative data are available. The CBCL has high retest reliability, interparent agreement, and validity. It was highly correlated with similar parent measures of child behavior, and scaled scores and clinical cutpoints discriminated between referred and nonreferred children.
Change in Child Behavior Checklist (CBCL) - total externalizing score | Change from pre-treatment to post-treatment (an average of 16 weeks)
  The CBCL (Achenbach, 2001) is a 118-item parent-report scale assessing behavioral problems and social competencies. Only parents will complete this measure. Items are rated from not true (0) to very true or often true (2). The CBCL has broadband internalizing and externalizing factors and eight specific scales (e;g., anxiety-depression). Normative data are available. The CBCL has high retest reliability, interparent agreement, and validity. It was highly correlated with similar parent measures of child behavior, and scaled scores and clinical cutpoints discriminated between referred and nonreferred children.
Change in Responses to Stress Questionnaire (RSQ)-Youth | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The RSQ (Connor-Smith et al., 2000) will be used to assess youth-self-reports and parent-reports of the use of primary control and secondary control coping strategies in response to significant life stressors. Research with three samples of adolescents and two samples of parents (reporting on their adolescents) has shown good evidence for the psychometric integrity of the measure. The factor structure of the RSQ has been tested and replicated using confirmatory factor analysis across three stressor classes in two samples. And both internal consistency and retest reliability of the five factors are strong, across samples. Across samples, scores on the primary and secondary control coping factors have shown strong negative correlations with both internalizing and externalizing problems. The parent form consists of 68 items and can be administered to target anxiety (RSQP-Scared) or depressive feelings (RSQP-Bad). The child form (Responses to Stress) is a shorter 30-item scale.
Change in Responses to Stress Questionnaire (RSQ)- Parent | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The RSQ (Connor-Smith et al., 2000) will be used to assess youth-self-reports and parent-reports of the use of primary control and secondary control coping strategies in response to significant life stressors. Research with three samples of adolescents and two samples of parents (reporting on their adolescents) has shown good evidence for the psychometric integrity of the measure. The factor structure of the RSQ has been tested and replicated using confirmatory factor analysis across three stressor classes in two samples. And both internal consistency and retest reliability of the five factors are strong, across samples. Across samples, scores on the primary and secondary control coping factors have shown strong negative correlations with both internalizing and externalizing problems. The parent form consists of 68 items and can be administered to target anxiety (RSQP-Scared) or depressive feelings (RSQP-Bad). The child form (Responses to Stress) is a shorter 30-item scale.
Change in Behavioral Activation for Depression Scale - Adolescent (BADS-A); youth | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The BADS-Y is a 26-item adaptation of the adult BADS (Kanter et al., 1997; Kanter et al., 1999), rated on a "0" (Not at All) to "6" (Completely) scale, designed to assess level of behavioral activation and avoidance. Factor analysis in the adult version detected four factors: Activation, Avoidance/Rumination, Work/School Impairment, and Social Impairment) with good factor structure, internal consistency and test-retest reliability. Normative data was also collected in an adult community sample. BADS-A was adapted for the current study to reflect developmentally appropriate reading level and concepts.
Change in Behavioral Activation for Depression Scale - Adolescent (BADS-A); parent forms | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The BADS-Y is a 26-item adaptation of the adult BADS (Kanter et al., 1997; Kanter et al., 1999), rated on a "0" (Not at All) to "6" (Completely) scale, designed to assess level of behavioral activation and avoidance. Factor analysis in the adult version detected four factors: Activation, Avoidance/Rumination, Work/School Impairment, and Social Impairment) with good factor structure, internal consistency and test-retest reliability. Normative data was also collected in an adult community sample. BADS-A was adapted for the current study to reflect developmentally appropriate reading level and concepts.
Change in Child Automatic Thoughts Scale: child report | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  CATS (Schniering & Rapee, 2002) is a 40-item child-report measure designed to assess negative self-statements in children and adolescents. The CATS was developed and validated on a wide age range of youth (7 - 16 years old) and found to effectively discriminate between non-clinical youth and those with clinical anxiety, depression, and behavior disorders. Confirmatory factor analyses supported four distinct but strongly correlated factors relating to automatic thoughts on physical threat, social threat, personal failure and hostility. The internal consistency of the total score and subscales was high (α > .85) and test-retest reliability at 1 and 3 months was acceptable (r = .91).
Change in Affect and Arousal Scale: child report | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  AFARS (Chorpita, Daleiden, Moffitt, Yim, & Umemoto, 2000) is a 27-item child-report measure that assesses affective dimensions related to anxiety and depression. Consistent with the Tripartite theory of internalizing disorders, factor analysis of large, multi-ethnic samples support a three factor structure of Negative Affect, Positive Affect, and Physiological Hyperarousal. Validation studies have provided preliminary evidence of acceptable 1-week test-retest reliability, convergent validity, and discriminant validity for the AFARS PA, NA, and PH scales Daleiden, CHorpita, & Lu, 2000).
Change in Difficulties in Emotion Regulation Scale: child report | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  DERS (Gratz & Roemer, 2004) is a 41-item measure evaluating six domains of emotion regulation, including: (1) Nonacceptance of Emotional Reponses (Non-acceptance), (2) Difficulties Engaging in Goal-Directed Behavior (Goals), (3) Impulse Control Difficulties (Impulse), (4) Lack of Emotional Awareness (Awareness), (5) Limited Access to Emotion Regulation Strategies (Strategies), and (6) Lack of Emotional Clarity (Clarity). The Difficulties Engaging in Goal-Directed Behavior subscale is most conceptually related to distress tolerance. The DERS has demonstrated good test-retest reliability over a period of 4-8 weeks (r = 0.88, p < .01), adequate internal consistency for each subscale (α > .80), and high internal consistency (α = 0.93). Items are rated on a 5-point scale ranging from (1) almost never to (5) almost always, with higher scores indicating greater emotion dysregulation.
Change in Real-time Emotion Action and Cognition Tracker (REACT) system: child | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The REACT system (Chu, Skriner, Silk, & Nock, 2009) is an electronic diary system that can be completed by a respondent on a smart phone, ipod, or computer via a website. The 169 screen interview is administered through the Symtrend mobile application (https://www.symtrend.com/) which provides a customizable interface for creating electronic diary interviews. REACT will be used to evaluate relations between mood and coping at three points in treatment (intake, midtreatment, and posttreatment). It has been piloted with 53 youth (ages 12-14 years old; Chu, Crocco, Esseling, Areizaga, Lindner, & Skriner, 2016) and reliably distinguished non-clinical youth from anxious/depressed youth in frequency of behavioral disengagement and intensity of emotions experienced.
Change in Rearing Behaviors Questionnaire: child | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The Rearing Behaviors Questionnaire is a 33-item instrument designed to capture three aspects of parenting behavior: Psychological Control, Autonomy versus Overprotection, and Acceptance versus Rejection. The RBQ combines the 23-item Mother-Father-Peer Inventory (MFP; Epstein, 1983) with the 10-item Psychological Control subscale of the Child Report of Parental Behavior Inventory (CRPBI; Schludermann & Schludermann, 1970), creating a measure that taps parenting constructs reflective of etiological models of anxiety disorders in children.
Change in Rearing Behaviors Questionnaire: parent | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The Rearing Behaviors Questionnaire is a 33-item instrument designed to capture three aspects of parenting behavior: Psychological Control, Autonomy versus Overprotection, and Acceptance versus Rejection. The RBQ combines the 23-item Mother-Father-Peer Inventory (MFP; Epstein, 1983) with the 10-item Psychological Control subscale of the Child Report of Parental Behavior Inventory (CRPBI; Schludermann & Schludermann, 1970), creating a measure that taps parenting constructs reflective of etiological models of anxiety disorders in children.
Change in Family Environment Scale - parent and child | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  is a 90-item multi-respondent (parent/child) scale that measures each member's perspective on family environment. Four of the 10 subscales (36 items) will be used to assess control (degree of set rules and procedures used to run the family), cohesion (degree of commitment to help and support family members), independence (extent to which family members are assertive and self sufficient), and conflict (amount of openly expressed anger and conflict). The FES is the most widely used measure of family climate with well-documented reliability and validity (Moos & Moos, 2009). The four chosen subscales have also been most consistently associated with internalizing (anxiety/depression) problems in youth. Respondents complete 36 True/False statements about their families; lower scores equate to more negative family environments.
Change in Me and My Mother (MMM): child report | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The MMF and the MMM (Wood, Kiff, & Piacentini, 2005) are 33-item child-report scales designed to assess the child's perspective of concrete, observable parent-child interactions that have occurred during a 1-week timeframe. The two companion scales allow the child to report on interactions with both father and mother. Items focus on (a) parents providing help with private daily routines that most school-age children are capable of performing independently (e.g., dressing, bathing), (b) intrusions on children's personal space (lying with child on his/her bed at night), and (c) infantilizing behavior (e.g., using baby words).
Change in Me and My Father (MMF): child report | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The MMF and the MMM (Wood, Kiff, & Piacentini, 2005) are 33-item child-report scales designed to assess the child's perspective of concrete, observable parent-child interactions that have occurred during a 1-week timeframe. The two companion scales allow the child to report on interactions with both father and mother. Items focus on (a) parents providing help with private daily routines that most school-age children are capable of performing independently (e.g., dressing, bathing), (b) intrusions on children's personal space (lying with child on his/her bed at night), and (c) infantilizing behavior (e.g., using baby words).
Change in Depression Anxiety Stress Scales-21 (DASS-21) - parent | Change from pre-treatment to post-treatment (an average of 16 weeks)
  The DASS-21 is a widely used self-report measure that assesses symptoms of anxiety, stress, and depression in adults. Parents will complete this measure about themselves. The DASS-21 will be used to assess the parent's own symptom and stress levels. It asks respondents to indicate the extent to which each item was applicable over the previous week using a 0-3 scale with the following response options: did not apply to me (0), applied to me to some degree, or some of the time (1), applied to me a considerable degree, or a good part of the time (2), applied to me very much, or most of the time (3). The DASS-21 distinguishes well between features of depression, physiological arousal, and psychological tension (Antony, Beiling, Cox, Enns, & Swinson, 1998), and has scores in the acceptable to excellent ranges. Additionally, the measure has been demonstrated to be a valid tool for assessing client outcomes in routine clinical practice (Ng, Trauer, Dodd, Callaly, Campbell, & Berk, 2007).
Change in Parent-Child Interaction Questionnaire (PCIQ) - parent report | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The PCIQ (Wood, Kiff, & Piacentini, 2005) is the parent-report version of the MMF and MMM parent-child interaction scales. The parent version uses a rating scale that is based on the frequency of each behavior: 1 (This never or almost never occurred [0-1 days this week]), 2 (This sometimes occurred [2-5 days this week]), or 3 (This almost always occurred [6-7 days this week]).
Change in Parental Acceptance and Action Questionnaire (PAAQ) - parent report | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  PAAQ (Cheron, Ehrenreich, & Pincus, 2009). The PAAQ is a 15-item questionnaire based on Hayes' Acceptance and Action Questionnaire (2004), but modified to assess experiential avoidance specifically in the context of parenting. Parents report attitudes toward their child's distress on a Likert-type scale ranging from Never True (1) to Always True (7). The PAAQ is comprised of two factors, Unwillingness (parents' unwillingness to witness their child experience negative emotion) and Inaction (parents' inability to effectively manage their reactions to their child's affect). Psychometric data indicate moderate test-retest reliability, r=.72, and support the temporal stability, internal consistency, and criterion validity of the measure.
Change in Stroop Color-Word Association Test error score: child | Change from pre-treatment to post-treatment (an average of 16 weeks)
  SCWT (Stroop, 1935), used with children 6 years and older, assesses selective attention, response inhibition, and controlled cognitive processing. In its standard format (Golden, 1978), the SCWT features three subtests: Stroop Word (SW), Stroop Color (SC), and Stroop Color-Word (SCW). All three Stroop subtests comprise 100 items and scoring is based on the number of items read or named correctly within a 45-second time interval. All three subtests have demonstrated good test-retest reliability (r > 0.80; Connor, Franzen, & Sharp, 1988; Graf, Utte, & Tuokko, 1995).
Change in Emotional Stroop error score: child | Change from pre-treatment to post-treatment (an average of 16 weeks)
  ES (Weissman, 2007; adapted from Taghavi et al., 2003) features four subtests each comprising twelve words categorized threat-related, depression-related, happy, or neutral. The format and administration of the four modified Stroop subtests match the standard SCWT, and the order of the words were randomly generated for the current study. The adapted Stroop task used in the current investigation does not have well-documented psychometric properties. However, studies using a similar task have reported large effect sizes for anxiety-control group comparisons for threat versus neutral words (e.g., Taghavi et al., 2003; Cohen's d=.79)
Change in Therapeutic Alliance Scale for Children/Adolescents - therapist report | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The TASC and TASA (Shirk & Saiz, 1992) assess quality of youths' working alliance with their therapists. The 12-item scale comes in both a youth-report form and a parent-report form (parents reporting on their youth's relationship with the therapist). The youth measure has shown good internal consistency in a sample of 44 clinic-referred youth (alpha = .84), and good 7-14-day test-retest reliability (r=.65) in a sample of 16 clinic-referred youth. The parent measure has also shown good internal consistency in a sample of 47 parents of clinic-referred youth (alpha=.92), and good 7-14-day test-retest reliability (r=.82) in a sample of 25 parents of clinic-referred youth.
Change in Therapeutic Alliance Scale for Children/Adolescents - child | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The TASC and TASA (Shirk & Saiz, 1992) assess quality of youths' working alliance with their therapists. The 12-item scale comes in both a youth-report form and a parent-report form (parents reporting on their youth's relationship with the therapist). The youth measure has shown good internal consistency in a sample of 44 clinic-referred youth (alpha = .84), and good 7-14-day test-retest reliability (r=.65) in a sample of 16 clinic-referred youth. The parent measure has also shown good internal consistency in a sample of 47 parents of clinic-referred youth (alpha=.92), and good 7-14-day test-retest reliability (r=.82) in a sample of 25 parents of clinic-referred youth.
Change in Child Involvement Rating Scale-Therapist report | Trajectory of change every four weeks from pretreatment to postreatment (an average of 16 weeks)
  The CIRS (Chu & Kendall, 2004) is a 10-item child involvement rating scale originally designed as an observational coding scale. The therapist-report version (CIRS-T) allows the therapist to provide the therapist's perspective on child engagement each session. Six items assess examples of positive child engagement and four items assess negative child engagement. The CIRS has demonstrated strong internal consistency (coefficient alpha = .73), good re-test reliability (ICC= .59), and strong inter-rater reliability (ICC= .76) (Chu & Kendall, 2004).
Change in Service Assessment for Children and Adolescents (SACA) - Service Use Scale: parent report | Change from pre-treatment to post-treatment (an average of 16 weeks)
  An important question to ask about any treatment program is whether it reduces the need for other services. To address this question for the VGTS, we rely on the SACA (Horwitz et al., 2001), a standardized interview for parents, tapping use of mental health services across a broad spectrum (including outpatient, inpatient, and school-based). SACA reliability and validity data are now well-documented (Hoagwood et al., 2000; Horwitz et al., 2001; Stiffman et al., 2000).

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Chu, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Rutgers University (Youth Anxiety and Depression Clinic), Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
There is no intention to share IPD.

REFERENCES:
- [Background] Achenbach, T. M. (2001). Manual for the ASEBA Child Behavior Checklist for Ages 6-18. Burlington, VT: Achenbach System of Empirically Based Assessment.
- [Background] Chorpita BF, Yim L, Moffitt C, Umemoto LA, Francis SE. Assessment of symptoms of DSM-IV anxiety and depression in children: a revised child anxiety and depression scale. Behav Res Ther. 2000 Aug;38(8):835-55. doi: 10.1016/s0005-7967(99)00130-8. PMID 10937431
- [Background] Chorpita, B.F., Daleiden, E. L., Moffitt, C., Yim, L., & Umemoto, L. A. (2000). Assessment of tripartite factors of emotion in childrean and adolescent: I. Structural validity and normative data of an affect and arousal scale. Journal of Psychopathology and Behavioral Assessment, 22, 141-160.
- [Background] Connor-Smith JK, Compas BE, Wadsworth ME, Thomsen AH, Saltzman H. Responses to stress in adolescence: measurement of coping and involuntary stress responses. J Consult Clin Psychol. 2000 Dec;68(6):976-92. PMID 11142550
- [Background] Guy, W. (1976). ECDEU Assessment Manual for Psychopharmacology (2nd ed.) (DHEW Publication ABM 76-388). Washington, DC: US Government Printing Office.
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Graf P, Uttl B, Tuokko H. Color- and picture-word Stroop tests: performance changes in old age. J Clin Exp Neuropsychol. 1995 May;17(3):390-415. doi: 10.1080/01688639508405132. PMID 7650102
- [Background] Hoagwood, K., Horwitz, S., Stiffman, A., Weisz et al. (2000). Concordance between parent reports of children's mental health services and service records: The Services Assessment for Children and Adolescents. Journal of Child and Family Studies, 9, 315-331.
- [Background] Horwitz SM, Hoagwood K, Stiffman AR, Summerfeld T, Weisz JR, Costello EJ, Rost K, Bean DL, Cottler L, Leaf PJ, Roper M, Norquist G. Reliability of the services assessment for children and adolescents. Psychiatr Serv. 2001 Aug;52(8):1088-94. doi: 10.1176/appi.ps.52.8.1088. PMID 11474056
- [Background] Hodges, K. (1990). Depression and anxiety in children: A comparison of self-report questionnaires to clinical interview. Psychological Assessment, 2, 376-381.
- [Background] Kanter, J. W., Mulick, P. S., Busch, A. M., Berlin, K. S., & Martell, C. R. (1997). The Behavioral Activation for Depression Scale (BADS): Psychometric properties and factor structure. Journal of Psychopathology Behavioral Assessment, 29, 191-202.
- [Background] Kanter, J. W., Rusch, L. C., Busch, A. M.,& Sedivy, S. K. (1999). Validation of the Behavioral Activation for Depression Scale (BADS) in a community sample with elevated depressive symptoms. Journal of Psychopathology Behavioral Assessment, 31, 36-42.
- [Background] Kazdin, A. E. (1992). Research Design in Clinical Psychology, 2nd Ed. Needham Heights, MA: Allyn & Bacon.
- [Background] Kendall, P. (2000). Cognitive-behavioral therapy for anxious children: Therapist Manual (2nd ed.). Ardmore, PA: Workbook Publishing, Inc.
- [Background] March, J. S. (1997). Multidimensional Anxiety Scale for Children: Technical Manual. North Tonawanda, NY: Multi-Health Systems, Inc.
- [Background] Muris, P. (2001) A brief questionnaire for measuring self-efficacy in youths. Journal of Psychopathology and Behavioral Assessment. Vol 23(3), 145-149.
- [Background] Poznanski, E. O., Mokros, H.B. (1996). Manual for the Children's Depression Rating Scale-Revised. Los Angeles: Western Psychological Services.
- [Background] Radloff, L.S. (1977). The CES-D Scale: a self-report depression scale for research in the general population. Applied Psychological Measures, 1, 385-401.
- [Background] Richards A, Richards LC, McGeeney A. Anxiety-related Stroop interference in adolescents. J Gen Psychol. 2000 Jul;127(3):327-33. doi: 10.1080/00221300009598587. PMID 10975428
- [Background] Schniering CA, Rapee RM. Development and validation of a measure of children's automatic thoughts: the children's automatic thoughts scale. Behav Res Ther. 2002 Sep;40(9):1091-109. doi: 10.1016/s0005-7967(02)00022-0. PMID 12296494
- [Background] Shirk, S., & Saiz, C. (1992). Clinical, empirical, and developmental perspectives on the therapeutic relationship in child psychotherapy. Development and Psychopathology, 4, 713-728.
- [Background] Silverman, W. K., & Albano, A. A. (1996). Anxiety Disorders Interview Schedule (ADIS-IV) Child and Parent Interview Schedules. US: Graywind Publications.
- [Background] Silverman WK, Nelles WB. The Anxiety Disorders Interview Schedule for Children. J Am Acad Child Adolesc Psychiatry. 1988 Nov;27(6):772-8. doi: 10.1097/00004583-198811000-00019. No abstract available. PMID 3198566
- [Background] Spielberger, C. (1973). State-Trait Anxiety Interview for Children: Professional Manual. Redwood City, CA: Mind Garden, Inc.
- [Background] Stiffman AR, Horwitz SM, Hoagwood K, Compton W 3rd, Cottler L, Bean DL, Narrow WE, Weisz JR. The Service Assessment for Children and Adolescents (SACA): adult and child reports. J Am Acad Child Adolesc Psychiatry. 2000 Aug;39(8):1032-9. doi: 10.1097/00004583-200008000-00019. PMID 10939232
- [Background] Strauss, C. (1987). Modification of trait portion of State-Trait Anxiety Inventory for Children-parent form. (Available from the author, Department of Psychology, University of Florida, Gainesville, FL 32606)
- [Background] Stroop, J. (1935). Studies of interference in serial verbal reactions. Journal of Experimental Psychology, 28, 643-662.
- [Background] Weisz JR, Thurber CA, Sweeney L, Proffitt VD, LeGagnoux GL. Brief treatment of mild-to-moderate child depression using primary and secondary control enhancement training. J Consult Clin Psychol. 1997 Aug;65(4):703-7. doi: 10.1037//0022-006x.65.4.703. PMID 9256573